CLINICAL TRIAL: NCT04906668
Title: Pulmonary-vein Isolation or Ablation of Atrioventricular-node and Pacemaker Implantation for Elderly Patients With Persistent Atrial Fibrillation (ABLATE Versus PACE)
Brief Title: ABLATE Versus PACE: PVI or AV Node Ablation and PM Implantation for Elderly Patients With Persistent AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Josefs-Hospital Wiesbaden GmbH (Other)
Collaborators: The German Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABLATE versus PACE
Record Dates: First submitted 2021-05-19; First posted 2021-05-28 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoballoon pulmonary-vein isolation (Active Comparator)
  Interventions: Procedure: Cryoballoon pulmonary-vein isolation
- Ablation of atrioventricular-node and pacemaker implantation (Active Comparator)
  Interventions: Procedure: Pacemaker implantation and ablation of atrioventricular-node

INTERVENTIONS:
Procedure: Cryoballoon pulmonary-vein isolation — Electrical isolation of the pulmonary-veins using cryoenergy
  Arms: Cryoballoon pulmonary-vein isolation
Procedure: Pacemaker implantation and ablation of atrioventricular-node — Pacemaker implantation and ablation of atrioventricular-node
  Arms: Ablation of atrioventricular-node and pacemaker implantation

SUMMARY:
As patients age, symptom control and treatment of atrial fibrillation become equally difficult, often leading to increased hospitalization. ABLATE versus PACE is a prospective, randomized clinical trial comparing pacemaker implantation with AV node ablation with pulmonary vein isolation in terms of rehospitalization and quality of life in patients with persistent AF aged 75 years and older.

DETAILED DESCRIPTION:
Atrial fibrillation is the most common cardiac arrhythmia and is a major public and represents a major public health problem with increasing healthcare costs and increased mortality risk.

In case of recurrent symptomatic atrial fibrillation current guidelines recommend pulmonary-vein isolation (PVI) as invasive treatment option. However, 5-year arrhythmia-free survival estimate is 29% after single catheter ablation. Although the long-term success rates in maintaining sinus rhythm are higher than with drug-based rhythm control, they are still moderate, especially in older patients with comorbidities. Therefore, repeated interventions are often necessary.

An effective method for frequency control is atrioventricular (AV) node ablation after implantation of a pacemaker ("ablate-and-pace"). In this case, the ventricular rate is only set by the pacemaker and can be programmed according to the patient's needs.

There are some theoretical disadvantages of this treatment option (pacemaker dependency, reduction of cardiac outpout due to lack of atrial contraction) which is why this method nowadays is almost exclusively used in older (and physically less active) patients.

The ABLATE versus PACE trial is a prospective randomized clinical trial comparing at 196 these two treatment options in terms of rehospitalizations due to cardiovascular causes and quality of life in elderly patients (≥ 75 years) with normal ejection fraction (≥ 50%).

ELIGIBILITY:
Inclusion Criteria:

* Persistent AF according to current ESC guideline (2020)
* Symptoms EHRA classification II - IV despite guideline indicated medical therapy
* Age ≥ 75 years
* Capability of giving written informed consent

Exclusion Criteria:

* impaired systolic left ventricular function (ejection fraction < 50%)
* High-grade (III°) left cardiac valvular disease
* pre-implanted pacemaker
* bradycardia-indication for pacemaker
* Surgical coronary revascularization (within the last 90 days) or current triple therapy after stent PCI
* contraindication for PVI or pacemaker-implantation
* contraindication for oral anticoagulation
* body-mass-index BMI > 40 kg/m2
* inability to give written informed consent
* concomitant participation in another registered trial
* life expectancy < 12 months
* reversible cause of AF (e.g. thyrotoxicosis, alcohol ingestion)

Ages: 75 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with any hospitalization due to atrial fibrillation, atrial tachycardia or flutter after blanking period or cardiac decompensation requiring inpatient treatment | 36 months
  except for protocol-indicated AVN ablation
Number of subjects requiring repeat ablation, electrical or pharmacological cardioversion for symptomatic relapse of atrial fibrillation, atrial tachycardia or flutter after blanking period | 36 months
Number of subjects requiring upgrade to cardiac resynchronization therapy pacemaker due to reduced systolic left ventricular function with ejection fraction ≤35% in "ablate-and-pace" group | 36 months

SECONDARY OUTCOMES:
Death from any cause | 36 months
Number of subjects with procedure-associated complications | 36 months
  (major bleeding by Bleeding Academic Research Consortium Definition (BARC ≥ 2) criteria, major groin site complications prolonging inpatient stay, pacemaker pocket bleeding prolonging inpatient stay, pericardial effusion, cerebrovascular or systemic embolism, phrenic nerve palsy, lead dislodgment, lead perforation, infection including pacemaker pocket infection, lead infection / pacemaker related endocarditis)
Number of subjects with nonfatal or fatal stroke/ transient ischemic attack (TIA) | 36 months
Quality of life as assessed by Atrial Fibrillation Effect on Quality-of-Life questionnaire (AFEQT) | 36 months
  Scale 20-140 with higher score indicating worse quality-of-life.
Deterioration of systolic LV function ≥10 percent | 36 months
Number of subjects requiring repeat ablation | 36 months
Number of subjects requiring anti-arrhythmic drug treatment after initial ablation | 36 months
Number of nights spent in hospital for occurrence of primary or secondary endpoints | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Ehrlich, MD, Principal Investigator — St. Josefs-Hospital Wiesbaden GmbH; Andreas Boehmer, MD, Principal Investigator — St. Josefs-Hospital Wiesbaden GmbH
Locations (12):
- Universitätsklinikum Innsbruck, Innsbruck, Austria
- Germany (11):
  - Kerckhoff-Klinik Bad Nauheim, Bad Nauheim
  - Vivantes Klinikum am Urban, Berlin
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt am Main, Frankfurt
  - Klinikum Fürth, Fürth
  - Ev. Krankenhaus Hagen-Haspe, Hagen
  - Asklepios Klinik St. Georg, Hamburg
  - Westpfalz-Klinikum Kaiserslautern, Kaiserslautern
  - Krankenhaus Landshut-Achdorf, Landshut
  - Universitätsklinikum Münster, Münster
  - St. Josefs-Hospital Wiesbaden GmbH, Wiesbaden

REFERENCES:
- [Background] Boehmer AA, Kaess BM, Ruckes C, Meyer C, Metzner A, Rillig A, Eckardt L, Nattel S, Ehrlich JR; ABLATE Versus PACE Investigators. Pulmonary Vein Isolation or Pace and Ablate in Elderly Patients With Persistent Atrial Fibrillation (ABLATE Versus PACE)-Rationale, Methods, and Design. Can J Cardiol. 2024 Dec;40(12):2429-2440. doi: 10.1016/j.cjca.2024.07.021. Epub 2024 Jul 25. PMID 39067619